CLINICAL TRIAL: NCT04894552
Title: Complications of Laparoscopic Hysterectomy and Sentinel Lymph Node Biopsy for Endometrial Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohammad Ahmed Magdy Abdelmonem Hussein Alzeiny, The principal investigator, Ain Shams Maternity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Hysterectomy and Sentinel LN
Record Dates: First submitted 2021-05-08; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Laparoscopic Hysterectomy and Sentinel Lymph Node Biopsy
Keywords: Endometrial carcinoma; Complications of Laparoscopic Hysterectomy; Sentinel Lymph Node Biopsy for Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: Patients with endometrial carcinoma will undergo laparoscopic hysterectomy and sentinel lymph node biopsy. The patient will be positioned in a modified lithotomy position with the hips flexed 30 degrees. Blue dye is injected at the cervix. The round ligament will be transected. Sentinel lymph nodes will be detected, dissected and isolated. Then standard lymphadenectomy will be done. Then the infundibulopelvic ligament will be transected. Ligation of the uterine vessels. The cardinal ligaments will be transected, and the vaginal fornices will be opened laparoscopically. The whole specimen will be removed through the vagina. The vaginal cuff will be then closed trans-vaginally. Intraoperative and early postoperative complications will be assessed. The isolated sentinel lymph node will be sent for pathological study as well as the standard lymphadenectomy specimens. Both specimens will be compared to assess the diagnostic reliability and sensitivity of the sentinel lymph node.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm clinical trial (Experimental): Convenience sampling method in which the first twenty cases of endometrial carcinoma patients who will undergo laparoscopic hysterectomy will be included. All cases will undergo laparoscopic hysterectomy. Sentinel lymph node biopsy will be detected, dissected and isolated. Then standard lymphadenectomy will be done
  Interventions: Procedure: Laparoscopic Hysterectomy and Sentinel Lymph Node Biopsy for Endometrial Carcinoma

INTERVENTIONS:
Procedure: Laparoscopic Hysterectomy and Sentinel Lymph Node Biopsy for Endometrial Carcinoma — Patients with endometrial carcinoma will undergo laparoscopic hysterectomy and sentinel lymph node biopsy. The patient will be positioned in a modified lithotomy position with the hips flexed 30 degrees. Blue dye is injected at the cervix. The round ligament will be transected. Sentinel lymph nodes will be detected, dissected and isolated. Then standard lymphadenectomy will be done. Then the infundibulopelvic ligament will be transected. Ligation of the uterine vessels. The cardinal ligaments will be transected, and the vaginal fornices will be opened laparoscopically. The whole specimen will be removed through the vagina. The vaginal cuff will be then closed trans-vaginally. Intraoperative and early postoperative complications will be assessed. The isolated sentinel lymph node will be sent for pathological study as well as the standard lymphadenectomy specimens. Both specimens will be compared to assess the diagnostic reliability and sensitivity of the sentinel lymph node.

SUMMARY:
Endometrial adenocarcinoma is believed to be a more treatable malignancy. Poor prognosis is associated with age, grade and depth of myometrial invasion, lymph node status, tumor size, invasion of lymphovascular space and involvement of the lower uterine segment. Sentinel lymph node (SLN) mapping can be considered as an al¬ternative to standard lymphadenectomy in the patients with apparently uterine-confined disease and to assess whether they have metastatic pelvic lymph nodes. Randomized trials, a Cochrane Database Systematic Review, and population-based surgical studies support minimally invasive techniques due to a lower rate of surgical site infection, ve¬nous thromboembolism, reduced hospitalisation, and lower cost of care. This is a one arm clinical trial pilot study that focuses on the intraoperative and early postoperative complications of laparoscopic hysterectomy in patients with endometrial carcinoma and assess the feasibility and the diagnostic reliability of sentinel lymph node biopsy.

DETAILED DESCRIPTION:
Patients with endometrial carcinoma will undergo laparoscopic hysterectomy and sentinel lymph node biopsy. The patient will be put under general anesthesia with endotracheal intubation. The patient will be positioned in a modified lithotomy position with the hips flexed 30 degrees. Patients will lie with legs open and slightly bent, with the buttocks protruding over the edge of the table. The patients' arms will be tucked at her sides. A Foley urinary catheter will be placed and Blue dye is injected at the cervix (2 ml at 3 o'clock and 2 ml at 9 o'clock (1 ml of the dye is injected deep and 1 ml is injected superficially)) and a uterine manipulator will be placed. The patient will be placed in the Trendlenburg position, and then pneumoperitoneum will be achieved through a Veress needle. Then four ports will be introduced (One 10 mm port at the umbilical incision, two 5 mm ports 4 cm medial and slightly above the level of the anterior superior iliac spines, and a 10 mm one midway between the umbilicus and the symphysis pubis). Blood vessels including the ovarian vessels and the uterine artery will be controlled by laparoscopic coagulating shears. After bowel manipulation out of the pelvis, the round ligament will be transected, and then the peritoneum over the psoas muscle will be cut lateral to the infundibulopelvic ligament, which will be retracted medially to permit identification of the iliac vessels and the ureter. The course of each pelvic ureter will be visualized through the medial leaf of the broad ligament. With medial traction on the utero-ovarian ligament or ovary, the peritoneal incision will be extended lateral to the ovarian vessels above the level of the pelvic brim to expose the area for lymphadenectomy. Sentinel lymph nodes will be detected, dissected and isolated. Then standard lymphadenectomy will be done. Then the infundibulopelvic ligament will be transected, care will be taken to ensure that the ureter will be secured. The anterior leaf of the broad ligament and anterior peritoneal reflection of the uterus will be opened. The bladder will be reflected anteriorly with atraumatic forceps introduced through the suprapubic sheath, and the bladder will be dissected from the cervix. Attention and care will be then directed to controlling the uterine artery lateral to the cervix. Care will be taken not to injury the ureter at this point. Ligation of the uterine artery and vein at their origin is preferred. The cardinal ligaments will be transected, and the anterior and posterior vaginal fornices will be opened laparoscopically and will be connected on both sides using the coagulation hook. The whole specimen will be removed through the vagina. The vaginal cuff will be then closed trans-vaginally by Vicryl sutures. Then the peritoneal cavity will be insufflated again and the laparoscope will be re-inserted to check for hemostasis before closure. Laparoscopic exit will be done after lavaging the operative field. Intraoperative and early postoperative complications will be assessed. The isolated sentinel lymph node will be sent for pathological study as well as the standard lymphadenectomy specimens. Both specimens will be compared to assess the diagnostic reliability and sensitivity of the sentinel lymph node.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have endometrial carcinoma and undergoing laparoscopic hysterectomy
* Estimated uterine upper margin is not beyond the midpoint between the umbilicus and the symphysis pubis.
* No preexisting cardiopulmonary dysfunction or poor control of systemic diseases.
* Bimanual pelvic examination confirmed good mobility of an enlarged uterus.
* Fractional curettage revealed no tumor extension in the endocervical canal.
* Preoperative metastatic work up revealed no extra-uterine disease either regional or systemic.

Exclusion Criteria:

* Patient refusal.
* Estimated uterine upper margin is beyond the midpoint between the umbilicus and the symphysis pubis.
* Cardiopulmonary dysfunction or poor control of systemic diseases.
* Bimanual pelvic examination confirmed fixed enlarged uterus.
* Fractional curettage revealed tumor extension in the endocervical canal.
* Preoperative metastatic work up revealed extra-uterine disease either regional or systemic.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications of laparoscopic hysterectomy in patients with endometrial carcinoma | one week
  To assess the intraoperative and early postoperative complications of laparoscopic hysterectomy in patients with endometrial carcinoma

SECONDARY OUTCOMES:
Sentinel lymph node biopsy operative time | one day
  The operative time for the sentinel lymph node biopsy and the operative time for the standard lymph adenectomy will be recorded and compared
Diagnostic reliability of sentinel lymph node biopsy in comparison to standard lymphadenectomy | one week
  Compare the histopathology reports of the sentinel lymph node biopsy and the standard lymphadenectomy as regards detection of malignant cells and record the number of times the sentinel lymph node biopsy missed the detetcion of malignant cells as compared to the standard lymphadenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elsenity, Prof., Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlin JN, Khoury-Collado F, Kim CH, Leitao MM Jr, Chi DS, Sonoda Y, Alektiar K, DeLair DF, Barakat RR, Abu-Rustum NR. The importance of applying a sentinel lymph node mapping algorithm in endometrial cancer staging: beyond removal of blue nodes. Gynecol Oncol. 2012 Jun;125(3):531-5. doi: 10.1016/j.ygyno.2012.02.021. Epub 2012 Feb 22. PMID 22366409
- [Background] Benedetti Panici P, Basile S, Salerno MG, Di Donato V, Marchetti C, Perniola G, Palagiano A, Perutelli A, Maneschi F, Lissoni AA, Signorelli M, Scambia G, Tateo S, Mangili G, Katsaros D, Campagnutta E, Donadello N, Greggi S, Melpignano M, Raspagliesi F, Cormio G, Grassi R, Franchi M, Giannarelli D, Fossati R, Torri V, Croce C, Mangioni C. Secondary analyses from a randomized clinical trial: age as the key prognostic factor in endometrial carcinoma. Am J Obstet Gynecol. 2014 Apr;210(4):363.e1-363.e10. doi: 10.1016/j.ajog.2013.12.025. Epub 2013 Dec 19. PMID 24361787
- [Background] Fader AN, Weise RM, Sinno AK, Tanner EJ 3rd, Borah BJ, Moriarty JP, Bristow RE, Makary MA, Pronovost PJ, Hutfless S, Dowdy SC. Utilization of Minimally Invasive Surgery in Endometrial Cancer Care: A Quality and Cost Disparity. Obstet Gynecol. 2016 Jan;127(1):91-100. doi: 10.1097/AOG.0000000000001180. PMID 26646127
- [Background] Holloway RW, Abu-Rustum NR, Backes FJ, Boggess JF, Gotlieb WH, Jeffrey Lowery W, Rossi EC, Tanner EJ, Wolsky RJ. Sentinel lymph node mapping and staging in endometrial cancer: A Society of Gynecologic Oncology literature review with consensus recommendations. Gynecol Oncol. 2017 Aug;146(2):405-415. doi: 10.1016/j.ygyno.2017.05.027. Epub 2017 May 28. PMID 28566221
- [Background] Janda M, Gebski V, Davies LC, Forder P, Brand A, Hogg R, Jobling TW, Land R, Manolitsas T, Nascimento M, Neesham D, Nicklin JL, Oehler MK, Otton G, Perrin L, Salfinger S, Hammond I, Leung Y, Sykes P, Ngan H, Garrett A, Laney M, Ng TY, Tam K, Chan K, Wrede CD, Pather S, Simcock B, Farrell R, Robertson G, Walker G, Armfield NR, Graves N, McCartney AJ, Obermair A. Effect of Total Laparoscopic Hysterectomy vs Total Abdominal Hysterectomy on Disease-Free Survival Among Women With Stage I Endometrial Cancer: A Randomized Clinical Trial. JAMA. 2017 Mar 28;317(12):1224-1233. doi: 10.1001/jama.2017.2068. PMID 28350928
- [Background] Koh WJ, Abu-Rustum NR, Bean S, Bradley K, Campos SM, Cho KR, Chon HS, Chu C, Cohn D, Crispens MA, Damast S, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, George S, Han E, Higgins S, Huh WK, Lurain JR 3rd, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Wyse E, Yashar CM, McMillian NR, Scavone JL. Uterine Neoplasms, Version 1.2018, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2018 Feb;16(2):170-199. doi: 10.6004/jnccn.2018.0006. PMID 29439178
- [Background] Mannschreck D, Matsuno RK, Moriarty JP, Borah BJ, Dowdy SC, Tanner EJ 3rd, Makary MA, Stone RL, Levinson KL, Temkin SM, Fader AN. Disparities in Surgical Care Among Women With Endometrial Cancer. Obstet Gynecol. 2016 Sep;128(3):526-34. doi: 10.1097/AOG.0000000000001567. PMID 27500330
- [Background] Scalici J, Laughlin BB, Finan MA, Wang B, Rocconi RP. The trend towards minimally invasive surgery (MIS) for endometrial cancer: an ACS-NSQIP evaluation of surgical outcomes. Gynecol Oncol. 2015 Mar;136(3):512-5. doi: 10.1016/j.ygyno.2014.11.014. Epub 2014 Nov 20. PMID 25462206
- [Background] Ueda SM, Kapp DS, Cheung MK, Shin JY, Osann K, Husain A, Teng NN, Berek JS, Chan JK. Trends in demographic and clinical characteristics in women diagnosed with corpus cancer and their potential impact on the increasing number of deaths. Am J Obstet Gynecol. 2008 Feb;198(2):218.e1-6. doi: 10.1016/j.ajog.2007.08.075. PMID 18226630